CLINICAL TRIAL: NCT06936306
Title: Effect of Professional Prophylaxis on Clinical Parameters and Patient Comfort: Randomized Slipt-Mouth Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lisbon (Other)
Collaborators: E.M.S. Electro Medical Systems S.A. (Unknown)
Responsible Party: Principal Investigator, João Nascimento, Principal Investigator, University of Lisbon
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: CE-FMDUL 202155
Record Dates: First submitted 2024-11-30; First posted 2025-04-20 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Dental Plaque; Gum Bleed
Keywords: Guided Biofilm Therapy; Dental plaque; Oral Hygiene; Air Polishing; Confort; Biofilm disclosing
MeSH Terms: conditions — Dental Plaque; Gingival Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test (Experimental): GBT Protocol
  Interventions: Procedure: GBT; Device: Master
- Control (Active Comparator): Scalling and polishing
  Interventions: Procedure: scalling

INTERVENTIONS:
Procedure: GBT — GBT Protocol
  Other Names: GBT Protocol
  Arms: Test
Device: Master — Use master piezon
  Arms: Test
Procedure: scalling — scalling
  Arms: Control

SUMMARY:
The goal of this clinical trial is to evaluate whether the Guided Biofilm Therapy (GBT) protocol can improve or maintain oral health and whether it provides more comfort to patients compared to a conventional protocol.

The study involved 25 adult patients aged 18 years or older, healthy, unmedicated, with more than 20 natural teeth, and no periodontitis.

Main Questions it Aims to Answer:

* Does the GBT protocol improve or maintain oral health compared to a conventional protocol?
* Is the GBT protocol more comfortable for patients than the conventional protocol? Comparison Group: Researchers compared the conventional protocol (used in quadrants I and III for Group A, and in quadrants II and IV for Group B) to the test GBT protocol (used in the opposite quadrants) to see if the GBT protocol results in improved clinical outcomes and better patient comfort.

Participants Will:

* Undergo two different protocols for oral prophylaxis (GBT and conventional protocols) on separate quadrants of their mouth.
* Have their clinical parameters assessed at three time points: baseline (T0), one week (T1), and three weeks (T2) after the intervention.
* Rate the comfort of the intervention using a Visual Analog Scale (VAS) on a Likert scale from 0 to 10 for each quadrant.

DETAILED DESCRIPTION:
After the initial evaluation of the participants and their inclusion in the study, the participants were randomized in blocks into group A where a conventional protocol was used in quadrants I and III and the test protocol in quadrants II and IV, and group B where a conventional protocol was used in quadrants II and IV and the test protocol in quadrants I and III.

The observations were made at three different times: baseline, one week after the intervention, and three weeks after the intervention. (Figure 1) The clinical assessment of each participant was performed using the the Ainamo & Bay gingival bleeding index (GBI), the O'Leary plaque control record (PCR) and the Silness and Löe plaque index (PI). (26-28) The primary outcome variable of the study was the Gingival Bleeding Index (GBI) with the Plaque Index (PI) as a secondary outcome variable.

Hard and soft deposits were removed according to the protocol assigned in one appointment performed by the principal investigator the day after the first data collection. The control protocol consisted of mechanical scaling with Woodpecker® scaler (Guilin, Guangxi, 541004 P.R.China) at power 1, followed by stain removal and polishing with R&S RUBBER DOME (R&S® Dental products 25, Rue Bleue - 75009 Paris) with Prophy Paste CCS® polishing paste RDA 250 (Directa AB P.O. Box 723, SE-194 27 Upplands Väsby, Sweden) at a speed of 10,000 rotations per minute.

The test protocol consisted in an assessment of the periodontal status following the application of the plaque discloser (Biofilm Discloser, Dr. Wittmann GmbH & Co KG 64673 Zwingenberg - Germany), followed by oral hygiene instructions and biofilm removal with an erythritol jet (Airflow Plus Powder®, Electro Medical Systems S.A.), Chemin de la Vuarpillière, 31, 1260 Nyon - Switzerland) with the Airflow Prophylaxis Master® device (Electro Medical Systems S.A., Chemin de la Vuarpillière, 31, 1260 Nyon - Switzerland). The jet stream was used at a power of 3 and the irrigation at a power of 10. Calculus removal was then performed with the piezon scaller of the same device using a PS scaler tip (Electro Medical Systems® S.A., Chemin de la Vuarpillière, 31, 1260 Nyon - Switzerland).

The first follow-up assessment (T1) was performed one week after the intervention, and the second follow-up assessment (T2) was performed 3 weeks after the intervention performed by the same research assistant that performed the initial assessment (T0). indecesThe precision and accuracy of the data collection was ensured by calibrating the instruments used and the investigators to minimize and control possible measurement errors. The assistant investigator underwent calibration before the start of the study to train the indeces, followed by a discussion of the criteria with the principal investigator.

After the appointment the participant rated comfort using a Visual Analog Scale measured on a Likert scale of 0 to 10 for each quadrant.

ELIGIBILITY:
Inclusion Criteria:

* healthy, unmedicated, without periodontitis, and with more than 20 natural teeth

Exclusion Criteria:

* dental implants, with periodontal pockets equal to or greater than 4, with fixed orthodontic appliances, with special needs, with some medical pathology, taking antibiotics 3 months before the study, smokers, with known hypersensitivity to erythritol and patients who did not complete the follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
GBI | 4 weeks
  Ainamo & Bay gingival bleeding index

SECONDARY OUTCOMES:
PCR | 4 weeks
  O'Leary plaque control record
PI | 4 weeks
  Silness and Löe plaque index

CONTACTS AND LOCATIONS:
Locations (1):
- University Lisbon, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/06/NCT06936306/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/06/NCT06936306/ICF_001.pdf